CLINICAL TRIAL: NCT04040426
Title: A Multi-center, Randomized Controlled ClinicalTrial Evaluating a Unique Bioactive SplitThickness Skin Allograft Versus Standard of Care in the Treatment of Diabetic Foot Ulcers
Brief Title: Bioactive Split Thickness Skin Allograft Versus Standard of Care in the Treatment of Diabetic Foot Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Professional Education and Research Institute (Other)
Collaborators: Solsys Medical LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOL-TRA-01
Record Dates: First submitted 2019-07-29; First posted 2019-07-31 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Diabetic Foot; Ulcer Foot
Keywords: Theraskin; Skin Graft; DFU; Ulcer
MeSH Terms: conditions — Diabetic Foot; Foot Ulcer; Ulcer

STUDY DESIGN:
Intervention Model Description: Multi-center, Randomized Controlled Clinical Trial Evaluating the Effect of Human Split Thickness Skin Graft Allograft (Theraskin™) in the Treatment of Diabetic Foot Ulcers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Human split thickness skin allograft (Theraskin™) (Experimental): Theraskin™ is an all-human split thickness skin allograft with a native extracellular matrix that can be used an adjunct to standard of care, for skin coverage in patients who have suffered from a diabetic foot wound in conjunction with offloading and Additional (outer) Dressing Application with moisture retention dressing. Theraskin™ is an allograft tissue and will be used in compliance with homologous use by the FDA under section 361 of the PHS Act and 21 CFR Part 1271
  Interventions: Other: Human split thickness skin allograft; Other: Additional Outer Dressing Applicaiton; Other: Offloading
- Fibracol wound dressing (Active Comparator): A commercially available wound dressing to be used per manufacturer's instructions for use on diabetic foot wounds in conjunction with offloading and Additional (outer) Dressing Application with moisture retention dressing moisture retention dressing
  Interventions: Other: Additional Outer Dressing Applicaiton; Other: Offloading; Other: Fibracol Wound Dressing

INTERVENTIONS:
Other: Human split thickness skin allograft — Application of a fenestrated human skin graft
  Other Names: Theraskin™
  Arms: Human split thickness skin allograft (Theraskin™)
Other: Additional Outer Dressing Applicaiton — Application of Moisture retentive dressing, and a multi-layer compression dressing
  Other Names: Outer protective dressing
Other: Offloading — Patient will be offloaded in a diabetic camboot after treatment, or total contact cast if patient cannot be fit with diabetic offloading boot
  Other Names: Pressure Relief
Other: Fibracol Wound Dressing — Application of Collagen Alginate Dressing
  Other Names: calcuim alginate
  Arms: Fibracol wound dressing

SUMMARY:
This study is a prospective, multi-center, randomized controlled trial designed to collect patient outcome data as well as assess performance and safety of a commercially available human split thickness skin allograft with SOC dressing compared to SOC dressings alone in the treatment of Diabetic Foot Wounds.

DETAILED DESCRIPTION:
This study is a prospective, multi-center, Randomized Controlled Trial ( RCT ) designed to assess performance and safety and collect patient outcome data on a commercially available human split thickness skin allograft (Theraskin™) with SOC dressing compared to SOC dressings alone in the treatment of Diabetic Foot Wounds (DFU) . The study will last thirteen weeks, with a two week screening period prior to enrollment. Theraskin™ is an allograft tissue and will be used in compliance with homologous use by the FDA under section 361 of the PHS Act and 21 CFR Part 1271.

There are two arms in the study:

Arm 1: The Experimental Arm , that will include SOC Therapy. SOC therapy in this study is offloading of the DFU (CAM boots or total contact casting [TCC] if the subject's foot is too large for a CAM), appropriate sharp or surgical debridement, infection management (systemic antibiotics only in conjunction with debridement) and application of human split thickness skin allograft (Theraskin™) followed by a moisture retention dressing and a padded 3-layer dressing comprised of 4x4 gauze pads, soft roll and compression wrap (DynaflexTM or equivalent).

Arm 2: The Standard of Care Arm. The SOC therapy in this study is offloading of the DFU (CAM boots or total contact casting [TCC] if the subject's foot is too large for a CAM), appropriate sharp or surgical debridement, infection management (systemic antibiotics only in conjunction with debridement) and wound care covering with calcium alginate Fibracol dressing followed by a moisture retentive dressing and a padded 3-layer dressing comprised of 4x4 gauze pads, soft roll and compressive wrap (DynaflexTM or equivalent).

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old.
* Presence of a DFU, Wagner Grade 1 (see Appendix A for definitions), extending at least through the dermis provided it is below the medial aspect of the malleolus.
* The index ulcer will be the largest ulcer if two or more DFUs are present with the same Wagner grade and will be the only one evaluated in the study. If other ulcerations are present on the same foot, they must be more than 2 cm distant from the index ulcer.
* Index ulcer (i.e. current episode of ulceration) has been present for greater than 4 weeks prior to SV1 and less than 1 year, as of the date the subject consents for study.
* Index ulcer is a minimum of 1.0 cm2 and a maximum of 25 cm2 at SV1 and TV1.
* Adequate circulation to the affected foot as documented by a dorsal transcutaneous oxygen measurement (TCOM) or a skin perfusion pressure (SPP) measurement of ≥ 30 mmHg, or an Ankle Branchial Index (ABI) between 0.7 and 1.3 within 3 months of SV1, using the affected study extremity. As an alternative arterial Doppler ultrasound can be performed evaluating for biphasic dorsalis pedis and posterior tibial vessels at the level of the ankle or a TBI (Toe Brachial Index) of > 0.6 is acceptable.
* The target ulcer has been offloaded for at least 14 days prior to randomization.
* Females of childbearing potential must be willing to use acceptable methods of contraception (birth control pills, barriers or abstinence) during the course of the study and undergo pregnancy tests.
* Subject understands and is willing to participate in the clinical study and can comply with weekly visits

Exclusion Criteria:

* Index ulcer(s) deemed by the investigator to be caused by a medical condition other than diabetes.
* Index ulcer, in the opinion of the investigator, is suspicious for cancer and should undergo an ulcer biopsy to rule out a carcinoma of the ulcer.
* Subjects with a history of more than two weeks of treatment with immune-suppressants (including systemic corticosteroids >10mg daily dose), cytotoxic chemotherapy, or application of topical steroids to the ulcer surface within 1-month prior to first SV1, or who receive such medications during the screening period or who are anticipated to require such medications during the course of the study.
* Subjects taking a selective COX-2 inhibitor, such as Celecoxib, for any condition.
* Subjects on any investigational drug(s) or therapeutic device(s) within 30 days preceding SV1.
* History of radiation at the ulcer site (regardless of time since last radiation treatment).
* Index ulcer has been previously treated or will need to be treated with any prohibited therapies.
* Presence of any condition(s) which seriously compromises the subject's ability to complete this study or has a known history of poor adherence with medical treatment.
* Osteomyelitis or bone infection of the affected foot as verified by x-ray within 30 days prior to randomization. (In the event of an ambiguous diagnosis, the Principal Investigator will make the final decision).
* Subject is pregnant or breast-feeding.
* Presence of diabetes with poor metabolic control as documented with an HbA1c >12.0 within last 90 days of randomization.
* Subjects with end stage renal disease as evidenced by a serum creatinine ≥3.0 mg/dL within 6 months of randomization.
* Index ulcer has reduced in area by 20% or more after 14 days of SOC from SV1 to the TV1/randomization visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-08-06 (Actual); Primary Completion 2021-09-14 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Percentage of index ulcers healed at 12 weeks | 12 weeks
  examine percent of ulcers healed at week twelve

SECONDARY OUTCOMES:
Percentage area reduction at 4 weeks | 4 weeks
  examine percent of wound reduction at 4 weeks
Percentage area reduction at 6 weeks | 6 weeks
  examine percent of wound reduction at 6 weeks
Percentage are reduction at 12 weeks | 12 weeks
  examine percent of wound reduction at 6 weeks
Percentage of index ulcers healed at 6 weeks | 6 weeks
  examine percent of ulcers healed at 6 weeks
Improvement in quality of life using Wound Quality of Life Score | 12 weeks
  The Wound-QoL, or wound quality of life questionnaire, measures the disease-specific, health-related quality of life of patients with chronic wounds. It consists of 17 items on impairments which are always assessed in retrospect to the preceding seven days. This questionnaire will be given to clinical trial participants at each visit, with the scale scores recorded. Each question is scored. Answers to each item are coded with numbers (0='not at all' to 4='very much'). As noted above the score will be reported with a minimam score of "0" and a maximum score of 68
Change in pain levels during trial, using the FACES pain scales which measure pain on a range of 0-10, zero being no pain and 10 being the most severe pain | 12 weeks
  The FACES pain scale will be administered to the clinical trial participants at each visit. The trial participant will select their pain level with a series of faces that correspond to a number between 0 which implies no pain , up to 10 which implies the most severe pain. The scores will be recorded for each clinical trial participant on each visit
Changes in peripheral neuropathy using Semmes Weinstein Monofilament "10"point | 12 weeks
  Each clinical trial participant will be examined by the principal investigator with a Semmes Weinstein monofilament wire at 10 points on the study foot, this standardized exam will be scored out of a total of 10 at each visit and recorded

CONTACTS AND LOCATIONS:
Overall Officials: Robert Galiano, MD, Principal Investigator — Northwestern University; David Armstrong, DPM, MD, PhD, Principal Investigator — USC Keck School of Medicine - Salsa
Locations (5):
- United States (5):
  - Center for Clinical Research, San Francisco, California
  - Gateway Clinical Trials LLC, O'Fallon, Illinois
  - Lower Extremity Institute of Research and Therapy, Youngstown, Ohio
  - Martinsville Research Institute, Martinsville, Virginia
  - Foot and Ankle Associates of Southwest VA, Salem, Virginia

IPD SHARING:
Plan to Share IPD: No